CLINICAL TRIAL: NCT00288418
Title: A Controlled, Randomized, Single-Blind, Multi-Center Pivotal Clinical Study Using Angiotech CVC to Prevent Bacterial Colonization on Short-Term Central Venous Catheters
Brief Title: Safety and Efficacy Study of Angiotech Central Venous Catheter to Prevent Bacterial Catheter Colonization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Angiotech Pharmaceuticals (Industry)
Responsible Party: Rui Avelar/ CMO, Angiotech
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 011-ACVC05
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Bacterial Infections
Keywords: Colonization of the catheter; Catheter related bloodstream infection
MeSH Terms: conditions — Bacterial Infections | interventions — Central Venous Catheters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARROWgard Blue® CVC (Active Comparator): 7-French x 20-cm, triple lumen, short-term CVC
  Interventions: Device: Central Venous Catheter
- Angiotech CVC (Experimental): A 7-French x 20-cm, triple lumen, short-term CVC with an anti-infective polymer coating, applied to the outer surface that contains the active pharmaceutical ingredient 5-fluorouracil (5-FU). The Angiotech CVC uses a 50µg/linear cm dose of 5-FU
  Interventions: Device: Central Venous Catheter

INTERVENTIONS:
Device: Central Venous Catheter — 7-French x 20-cm, triple lumen, short-term CVC vs. 7-French x 20-cm, triple lumen, short-term CVC with an anti-infective polymer coating, applied to the outer surface that contains the active pharmaceutical ingredient 5-fluorouracil (5-FU). The Angiotech CVC uses a 50µg/linear cm dose of 5-FU

SUMMARY:
The main purpose of this study is to determine if the Angiotech central venous catheter (CVC) is equal in effectiveness to a CVC coated with chlorhexidine and silver sulfadiazine in preventing bacterial catheter colonization. Other objectives of this study are to determine if the Angiotech CVC is equal in effectiveness to a CVC coated with chlorhexidine and silver sulfadiazine in preventing catheter-related local infection, and catheter-related bloodstream infection. This study will also assess the safety of the Angiotech CVC.

DETAILED DESCRIPTION:
Central venous catheters are widely used for hemodynamic monitoring and the administration of fluids, drugs, and nutrition. The most frequent life-threatening complication of central venous catheter use is septicemia. Normal cutaneous flora may invade the intracutaneous tract during or after catheter insertion. The colonizing bacteria subsequently disseminate along the catheter surface and ultimately seed into the blood stream.

In the United States, a total of 250,000 cases of central venous catheter-related infections are estimated annually. Costs per infection are estimated as high as US$56,000. It is clinically imperative that effective measures be found to decrease catheter infection rates while minimizing the risk of the development of microbial resistance.

Primary Objective: The primary objective of this study is to determine the non-inferiority of the Angiotech Central Venous Catheter (CVC) when compared to the ARROWgard Blue® CVC to prevent bacterial catheter colonization.

Secondary Objectives: The secondary objectives of this study are to determine the non-inferiority of the Angiotech CVC when compared to the ARROWgard Blue® CVC to prevent:

1. catheter-related local infection; and
2. catheter-related bloodstream infection.

Safety Objectives: This study will assess the safety of the Angiotech CVC.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* Be initially hospitalized in an intensive care setting
* Require insertion of a triple-lumen central venous catheter for an anticipated period of up to 28 days
* If female and of child-bearing potential, provide evidence of a negative pregnancy test

Exclusion Criteria:

* Has a life expectancy of less than one month
* Is pregnant
* Has a history of anaphylactic reactions, including reactions to contrast dyes
* Has a history of allergy to 5-fluorouracil (5-FU) or chlorhexidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Incidence of catheter colonization | Maximum of 28 days
  Primary Objective: The primary objective of this study was to determine the non-inferiority of the Angiotech Central Venous Catheter (CVC) when compared to the ARROWgard Blue® CVC to prevent bacterial catheter colonization.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Heard, MD, Principal Investigator — University of Mass. Medical School Department of Anesthesiology
Locations (21):
- United States (21):
  - Cardio-Thoracic Surgeons, P.C., Birmingham, Alabama
  - Pulmonary Consultant Group, Orange, California
  - Pulmonary Center Sharp Memorial Hospital, San Diego, California
  - Kaiser Permanente Santa Teresa, San Jose, California
  - Denver Health Medical Center, Denver, Colorado
  - Christiana Care Research Institute, Newark, Delaware
  - Florida Research Network, LLC, Gainesville, Florida
  - Atlanta Institute for Medical Research Inc, Decatur, Georgia
  - Kerry Thibodeaux, M.D., Opelousas, Louisiana
  - UMASS Medical School, Dept of Anesthesiology, Worcester, Massachusetts
  - Newark Beth Israel Hospital, Newark, New Jersey
  - Pulmonary and Critical Care Medicine, Cincinnati, Ohio
  - St Vincent Mercy Medical Center, Bldg 1, Toledo, Ohio
  - Medical University of Ohio, Toledo, Ohio
  - Universty of Oklahoma HSC, Oklahoma City, Oklahoma
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - University of Virginia, Department of Anesthesiology, Charlottesville, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Franciscan Health System Research Center, Tacoma, Washington